CLINICAL TRIAL: NCT04268303
Title: A Phase III Multicenter, Randomized, Double-Blind, Placebo-Controlled Study To Determine Efficacy and Safety of BXCL501 In Agitation Associated With Schizophrenia
Brief Title: Dexmedetomidine in the Treatment of Agitation Associated With Schizophrenia
Acronym: SERENITY I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioXcel Therapeutics Inc (Industry)
Collaborators: Cognitive Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BXCL501-301
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Results first posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Agitation; Schizophrenia; Schizo Affective Disorder; Schizoaffective Disorder; Schizophreniform Disorders
MeSH Terms: conditions — Psychomotor Agitation; Schizophrenia; Psychotic Disorders | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Phase III, Randomized, Double-Blind, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind, Placebo-Controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 120 Micrograms (Experimental): Sublingual film containing 120 Micrograms dexmedetomidine
  Interventions: Drug: Sublingual film containing dexmedetomidine (BXCL501)
- 180 Micrograms (Experimental): Sublingual film containing 180 Micrograms dexmedetomidine
  Interventions: Drug: Sublingual film containing dexmedetomidine (BXCL501)
- Placebo (Placebo Comparator): Sublingual placebo film
  Interventions: Drug: Placebo Film

INTERVENTIONS:
Drug: Sublingual film containing dexmedetomidine (BXCL501) — Sublingual film containing dexmedetomidine (BXCL501)
  Other Names: Dexmedetomidine
  Arms: 120 Micrograms; 180 Micrograms
Drug: Placebo Film — Placebo Film for BXCL501
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is a definitive study to support the safety and efficacy evaluation of BXCL501 for the acute treatment of agitation in schizophrenia. The BXCL501-301 study is designed to characterize the efficacy, safety and tolerability of BXCL501 (sublingual film formulation of DEX, HCl) in agitation associated with schizophrenia, schizoaffective disorder or schizophreniform disorder.

DETAILED DESCRIPTION:
The study will enroll approximately 375 subjects randomized 1:1:1 to dose regimens of 180µg, 120µg BXCL501, or placebo. Male and female adults with acute agitation associated with schizophrenia, schizoaffective disorder, or schizophreniform disorder will be enrolled. Eligible subjects may be identified in outpatient clinics, mental health, psychiatric or medical emergency services including medical/psychiatric observation units, or as newly admitted to a hospital setting for acute agitation or already in hospital for chronic underlying conditions. Subjects will be domiciled in a clinical research setting or hospitalized to remain under medical supervision while undergoing screening procedures to assess eligibility. Efficacy and safety assessments will be conducted periodically before and after dosing.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in the study if he or she meets the following criteria:

1. Male and female patients between the ages of 18 to 75 years, inclusive.
2. Patients who have met DSM-5 criteria for schizophrenia, schizoaffective, or schizophreniform disorder.
3. Patients who are judged to be clinically agitated at Screening and Baseline with a total score of ≥ 14 on the 5 items (poor impulse control, tension, hostility, uncooperativeness, and excitement) comprising the PANSS Excited Component (PEC).
4. Patients who have a score of ≥ 4 on at least 1 of the 5 items on the PEC at Baseline.
5. Patients who read, understand, and provide written informed consent.
6. Patients who are in good general health prior to study participation as determined by a detailed medical history, physical examination, 12-lead ECG with rhythm strip, blood chemistry profile, hematology, urinalysis, and in the opinion of the Principal Investigator.
7. Participants who agree to use a medically acceptable and effective birth control method

Exclusion Criteria:

A subject will be excluded from the study if he or she meets the following criteria:

1. Patients with agitation caused by acute intoxication, including positive identification of alcohol by breathalyzer or drugs of abuse (with the exception of THC) during urine screening.
2. Use of benzodiazepines, hypnotics and anti-psychotic drugs in the 4 hours before study treatment.
3. Treatment with alpha-1 noradrenergic blockers (terazosin, doxazosin, tamsulosin, alfuzosin, or prazosin) or other prohibited medications.
4. Patients who are judged to be at significant risk of suicide
5. Female patients who have a positive pregnancy test at screening or are breastfeeding.
6. Patients who have hydrocephalus, seizure disorder, or history of significant head trauma, stroke, transient ischemic attack, subarachnoid bleeding, brain tumor, encephalopathy, meningitis, Parkinson's disease or focal neurological findings.
7. History of syncope or other syncopal attacks, current evidence of hypovolemia, orthostatic hypotension.
8. Patients with laboratory or ECG abnormalities considered clinically significant by the investigator.
9. Patients with serious or unstable medical illnesses.
10. Patients who have received an investigational drug within 30 days prior to the current agitation episode.
11. Patients who are considered by the investigator, for any reason, to be an unsuitable candidate for receiving DEX.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Risinger, MD, Study Chair — BioXcel Therapeutics
Locations (15):
- United States (15):
  - BioXcel Clinical Research Site, Little Rock, Arkansas
  - BioXcel Clinical Research Site, Cerritos, California
  - BioXcel Clinical Research Site, Culver City, California
  - BioXcel Clinical Research Site, Long Beach, California
  - BioXcel Clinical Research Site, Orange, California
  - BioXcel Clinical Research Site, Miami Lakes, Florida
  - BioXcel Clinical Research Site, Chicago, Illinois
  - BioXcel Clinical Research Site, Gaithersburg, Maryland
  - BioXcel Clinical Research Site, Las Vegas, Nevada
  - BioXcel Clinical Research Site, Berlin, New Jersey
  - BioXcel Clinical Research Site, Marlton, New Jersey
  - BioXcel Clinical Research Site, Charleston, South Carolina
  - BioXcel Clinical Research Site, Austin, Texas
  - BioXcel Clinical Research Site, DeSoto, Texas
  - BioXcel Clinical Research Site, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Citrome L, Preskorn SH, Lauriello J, Krystal JH, Kakar R, Finman J, De Vivo M, Yocca FD, Risinger R, Rajachandran L. Sublingual Dexmedetomidine for the Treatment of Acute Agitation in Adults With Schizophrenia or Schizoaffective Disorder: A Randomized Placebo-Controlled Trial. J Clin Psychiatry. 2022 Oct 3;83(6):22m14447. doi: 10.4088/JCP.22m14447. PMID 36198061
- [Derived] Citrome L, Risinger R, Rajachandran L, Robison H. Sublingual Dexmedetomidine for Agitation Associated with Schizophrenia or Bipolar Disorder: A Post Hoc Analysis of Number Needed to Treat, Number Needed to Harm, and Likelihood to be Helped or Harmed. Adv Ther. 2022 Oct;39(10):4821-4835. doi: 10.1007/s12325-022-02274-3. Epub 2022 Aug 24. PMID 36002761
- See also: Journal Article — https://www.psychiatrist.com/jcp/schizophrenia/sublingual-dexmedetomidine-for-agitation-schizophrenia/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 120 Micrograms | 180 Micrograms | Placebo
Started | 129 | 125 (One participant enrolled in both the 120 microgram treatment group and subsequently the 180 microgram treatment group (at a second site) completed both courses of treatments, but is included only in the 120 microgram group for the randomized population.) | 126
Completed | 126 | 123 | 123
Not Completed | 3 | 2 | 3
Not completed — Lost to Follow-up | 1 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Adverse Event | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population (all participants who received study drug). One participant enrolled and randomized to the 120 μg group was enrolled a second time at a different site and randomized to the 180 μg group. The data from the first enrollment and treatment (120 μg) were included in the efficacy analyses. The data from both enrollments (120 μg and 180 μg) were included in the safety analyses and counted separately for each treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | 120 Micrograms | 180 Micrograms | Placebo | Total
Number analyzed (Participants) | 129 | 125 | 126 | 380
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (11.3) | 46.0 (11.9) | 45.1 (11.1) | 45.6 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 43 | 44 | 139
  Male | 77 | 82 | 82 | 241
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 13 | 7 | 37
  Not Hispanic or Latino | 112 | 112 | 119 | 343
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 92 | 102 | 102 | 296
  White | 33 | 21 | 21 | 75
  Other | 4 | 2 | 3 | 9
  Hispanic or Latino | 17 | 13 | 7 | 37
Positive and Negative Syndrome Scale-Excited Component [Mean (Standard Deviation); unit: units on a scale] — Population: One participant enrolled and randomized to the 120 μg group was enrolled a second time at a different site and randomized to the 180 μg group. The data from the first enrollment and treatment (120 μg) were included in the efficacy analyses. The data from both enrollments (120 μg and 180 μg) were included in the safety analyses and counted separately in each treatment group; they were counted once when dose groups were combined.
  units on a scale | 17.5 (2.5) | 17.6 (2.7) | 17.6 (2.3) | 17.6 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale- Excited Component (PEC) Total Score
Description: The Positive and Negative Syndrome Scale-Excited Component (PEC) includes 5 items-poor impulse control, tension, hostility, uncooperativeness, and excitement-each of which is rated from 1 (minimum) to 7 (maximum); the sum of these 5 items, the PEC total score, ranges from 5 (absence of agitation) to 35 (extremely severe).
Time Frame: Baseline and 2 hours
Population: Intent-to-Treat population, defined as all participants in the safety population who have a PEC score post-dose.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 120 Micrograms | 180 Micrograms | Placebo
Number analyzed (Participants) | 129 | 125 | 126
score on a scale
  Baseline | 17.5 (2.46) | 17.6 (2.69) | 17.6 (2.26)
  2 Hours | -8.4 (4.83) | -10.4 (4.34) | -4.7 (4.69)
Statistical Analysis 1: Comparison: 180 Micrograms vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: 120 Micrograms vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis

2. Secondary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale- Excited Component (PEC) Total Score Over Time
Description: Effect on agitation onset was measured by change from baseline in the Positive and Negative Syndrome Scale- Excited Component (PEC) total score. The Positive and Negative Syndrome Scale-Excited Component (PEC) includes 5 items-poor impulse control, tension, hostility, uncooperativeness, and excitement-each of which is rated from 1 (minimum) to 7 (maximum); the sum of these 5 items, the PEC total score, ranges from 5 (absence of agitation) to 35 (extremely severe).
Time Frame: Baseline and 10, 20, 30, 45, 60, 90 minutes post-dose
Population: Intent-to-Treat population, defined as all participants in the safety population who have a PEC score post-dose.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 120 Micrograms | 180 Micrograms | Placebo
Number analyzed (Participants) | 129 | 125 | 126
score on a scale
  Baseline | 17.5 (2.46) | 17.6 (2.69) | 17.6 (2.26)
  10 minutes | -1.3 (2.50) | -2.0 (3.19) | -1.3 (2.17)
  20 minutes | -2.8 (4.03) | -3.9 (4.54) | -2.5 (3.20)
  30 minutes | -4.4 (4.90) | -5.7 (5.27) | -3.1 (3.56)
  45 minutes | -5.7 (5.18) | -7.6 (5.32) | -3.6 (3.78)
  60 minutes | -6.9 (5.06) | -8.8 (4.96) | -4.1 (4.16)
  90 minutes | -8.0 (5.00) | -9.8 (4.60) | -4.6 (4.38)
Statistical Analysis 1: Comparison: 180 Micrograms vs Placebo; 180 Micrograms versus placebo; 90 minutes post-dose; Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: 120 Micrograms vs Placebo; 120 Micrograms versus placebo; 90 minutes post-dose; Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: 180 Micrograms vs Placebo; 180 Micrograms versus placebo; 60 minutes post-dose; Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 4: Comparison: 120 Micrograms vs Placebo; 120 Micrograms versus placebo; 60 minutes post-dose; Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 5: Comparison: 180 Micrograms vs Placebo; 180 Micrograms versus placebo; 45 minutes post-dose; Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 6: Comparison: 120 Micrograms vs Placebo; 120 Micrograms versus placebo; 45 minutes post-dose; Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 7: Comparison: 180 Micrograms vs Placebo; 180 Micrograms versus placebo; 30 minutes post-dose; Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 8: Comparison: 120 Micrograms vs Placebo; 120 Micrograms versus placebo; 30 minutes post-dose; Test type: Superiority; p = 0.0075, Mixed Models Analysis
Statistical Analysis 9: Comparison: 180 Micrograms vs Placebo; 180 Micrograms versus placebo; 20 minutes post-dose; Test type: Superiority; p = 0.0032, Mixed Models Analysis
Statistical Analysis 10: Comparison: 120 Micrograms vs Placebo; 120 Micrograms versus placebo; 20 minutes post-dose; Test type: Superiority; p = 0.4097, Mixed Models Analysis
Statistical Analysis 11: Comparison: 180 Micrograms vs Placebo; 180 Micrograms versus placebo; 10 minutes post-dose; Test type: Superiority; p = 0.0457, Mixed Models Analysis
Statistical Analysis 12: Comparison: 120 Micrograms vs Placebo; 120 Micrograms versus placebo; 10 minutes post-dose; Test type: Superiority; p = 0.9720, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 30 days
Description: Adverse Events: The Safety Population included all participants in the Randomized Population who received at least 1 dose of double-blind investigational product. One participant enrolled and randomized to the 120 μg group was enrolled a second time at a different site and randomized to the 180 μg group. The data from both enrollments (120 μg and 180 μg) were included in the safety analyses and counted separately in each treatment group; they were counted once when dose groups were combined.
Arm/Group | 120 Micrograms | 180 Micrograms | Placebo
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/126 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/129 | 0/126 | 0/126
Other Adverse Events (participants affected / at risk) | 51/129 | 47/126 | 19/126
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 120 Micrograms (N=129) | 180 Micrograms (N=126) | Placebo (N=126)
Dizziness (Nervous system disorders) | 3 | 8 | 1
Dry mouth (Gastrointestinal disorders) | 10 | 5 | 2
Headache (Nervous system disorders) | 6 | 4 | 6
Hypoesthesia oral (Nervous system disorders) | 5 | 7 | 0
Hypotension (Vascular disorders) | 8 | 5 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 7 | 0
Paresthesia oral (Nervous system disorders) | 5 | 3 | 1
Somnolence (Nervous system disorders) | 28 | 29 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/03/NCT04268303/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT04268303/SAP_001.pdf